CLINICAL TRIAL: NCT05356325
Title: The Role of FGF23 on the Induction of Cardiovascular Damage in Anemia With an Without Chronic Kidney Disease
Brief Title: FGF23 and Cardiovascular Damage in Anemia With an Without Chronic Kidney Disease.
Status: Recruiting | Type: Observational
Sponsor: Maimónides Biomedical Research Institute of Córdoba (Other)
Collaborators: Fondo de Investigacion Sanitaria (Other)
Responsible Party: Sponsor
Other Study IDs: PI20/1645
Record Dates: First submitted 2021-12-30; First posted 2022-05-02 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Fibroblast Growth Factor 23; Anemia; CKD
Keywords: FGF23; anemia; CKD; iron deficiency; cardiovascular risk; miRNAS; inflammation
MeSH Terms: conditions — Anemia; Iron Deficiencies; Inflammation

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples Without DNA — Blood samples Urine samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Anemia is associated with cardiovascular disease. Iron deficiency is usually induced in chronic kidney disease (CKD). In clinical studies, an inverse association between serum levels of iron and fibroblast growth factor 23 (FGF23), a cardiovascular risk factor, has been demonstrated. In addition, a number of the I.V. iron presentations mostly used to treat anemia show unwanted side effects related to phosphate alterations and increased FGF23. Objectives. The General Objective of this project is to evaluate, through in vivo and in vitro studies, the cardiovascular alterations related to the anemia-induced increase in FGF23 production; as well as the identification of possible molecular targets that may be useful in its prevention and/or palliation. Specific Objectives are: 1) To determine in a population with anemia (due to iron deficiency), with and without CKD, an association between the parameters related to iron metabolism, FGF23 and markers of cardiovascular damage. 2) To evaluate in vivo, in a murine experimental model of anemia, with and without CKD, the effects of the modulation (inhibition) of triggers of iron deficiency (hepcidin) and of the increase in FGF23 (HF1α), on markers of cardiovascular damage. 3) To compare in vivo, in an experimental model of anemia with and without CKD, the effect of different I.V. iron presentations (ferrous sulphate, ferric carboxymaltose and ferric citrate) on FGF23 levels and their cardiovascular impact. 4) To evaluate in vitro, in cardiomyocytes cultures, in the presence of iron deficiency, the direct effect of FGF23 on the induction of cardiac damage. 5) To evaluate in vitro, in osteoblasts cultures, the direct effect of ferrous sulphate, ferric carboxymaltose, ferric citrate and hepcidin. Methodology. The levels of intact and C-terminal FGF23 (FGF23i and FGF23c), the differential expression profile of plasma miRNAS and of proteomic, markers of cardiovascular disease, mineral metabolism, inflammation and oxidative stress and intracellular signalling pathways will be evaluated.

DETAILED DESCRIPTION:
1 Study populations 1.1) Study in patients with iron deficiency anemia with normal renal function. The study will be carried out in the serum samples of patients. All patients will be provided with the corresponding informed consent.

Patients with an age ≥18 years, normal renal function (GFR> 60 ml / min / 1.73m2), hemoglobin levels <11 g / dl, serum ferritin levels <100ng / dL or saturation percentage of transferrin <30%. Patients who have a history of treated or active malignancy, proliferative hematological disorders or evidence of malnutrition (BMI <17), who are receiving oral iron treatment, or who have had intestinal bleeding or have received a blood transfusion in the last 90 days, will be excluded from the study.

1.1.2) Study in patients with anemia and CKD. This study will include patients with stage 3 and 4 of kidney disease with or without anemia that meet the criteria: age ≥18 years, hemoglobin levels <11 g / dl, serum ferritin levels <100ng / dL or percentage Transferrin saturation <30%. Patients who have severe proteinuria, symptoms of treated or active malignancy, inflammatory rheumatic diseases, HIV positivity, Hepatitis B or C virus, who are receiving anticoagulation with coumarin or any erythropoiesis stimulating agent, who have undergone a major surgery or had a cardiovascular event, intestinal bleeding or received a blood transfusion in the last 3 months prior to the start of the study will be excluded.

In relation to the sample size required for the development of the study, it is considered that a random sample of 183 individuals for the population of patients with iron deficiency anemia without CKD and 218 for the study to be carried out with patients with anemia and CKD, will be enough to estimate, with a 95% confidence and an accuracy of +/- 5 percentage units, a population percentage that is expected to be around 13% and 15%, respectively. As a percentage of necessary replacements, it is expected to be 5% and 10%, respectively. 1.2. Determinations A blood simple will be taken at the initial time (before receiving treatment), 12 months after the start of iron supplementation, which will be ferrous sulfate or ferric carboxymaltose for patients. The blood sample will be centrifuged immediately at 3500 r.p.m for 10 'and stored at -80 ° C until the analysis of the different study parameters. The levels of Ca, creatinine, urea, phosphorus, albumin, hemoglobin, ferritin and iron saturation levels will be determined, using standardized and automated commercial assays (Beckman AU), which will be processed. The determination of intact and C-terminal FGF23 levels will be carried out by E.L.I.S.A. using the Kainos Laboratories kit, Japan and Immutopics, CA, respectively. For the analysis of PTH levels, the intact PTH Kit (Immutopics, CA) will be used. Hepcidin will be determined by ELISA (Elabsciences, USA).The levels of 25 (OH) D will be determined by radioimmunoassay (RIA) (Immunodiagnostic Systems, UK). Renal function will be performed by calculating the glomerular filtration rate (eGFR) using the CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration) formula, which includes serum creatinine, age, sex and race as variables. ELISA kits will be used for the quantitative determination of circulating levels of brain natriuretic peptide (BNP), myoglobin, and troponin, I, (Thermofisher scientific) and Bioplex to determine the levels of secreted cytokines. For the determination of oxidative stress in plasma, the activity of the enzyme glutathione peroxidase (GPX) will be analyzed, using the method of Flohé and Günzler.

Establishment, through the use of the latest technology of the non-coding transcriptomic profile (microRNAs) in the plasma of anemic patients without or with CKD and its association with the clinical and analytical profile of these pathologies. miRNAs profile study will be carried out with the Illumina SE50 platform (Novogene enterprise, Cambridge Science Park, UK). The study will be performed from plasma samples of patients with iron deficit and with or without renal failure. DEGseq R package will be used for identifying a differential expression. Gene Ontology (GO) enrichment analysis will be used on predicted target gene candidates of known and novel miRNAs. Kyoto Encyclopedia of Genes and Genomes (KEGG) pathway analysis will be used for identifying significantly enriched metabolic pathways or signal transduction pathways associated with differentially expressed miRNA target genes. A representative number of samples (n = 15 patients from each experimental situation including control subjects) will be considered. To validate the data obtained, real-time polymerase chain reaction (RT-PCR) of the selected miRNAS, differentially expressed, will be performed. The results obtained will be statistically analyzed to find possible correlations and associations with clinical and analytical parameters.

Proteomic analysis by mass spectrometry and its association with the clinical and analytical parameters of these pathologies. Mass spectrometry (MS) is an analytical technique in which the atoms or molecules of a sample are ionized, separated according to their mass/charge ratio (m/z) and subsequently detected and recorded. To carry out the proteomic study, the sera from the patient populations described above) will be depleted to eliminate the majority proteins. After a protein quantification, samples will be stored at -80 until the proteomic analysis is carried out. The sample will be treated appropriately and the tryptic peptides obtained will be analyzed by liquid nano-chromatography (reverse phase) coupled to mass spectrometry (nHPLC-MS) in order to quantify the relative abundance of proteins between the different conditions studied. For this, a mass spectrometer (Triple TOF 5600 + model, ABSciex) will be used working in the SWATH (Sequential Window Acquisition of all THeoretical Mass Spectra) acquisition mode. A representative number of samples (n = 15 patients from each experimental situation including control subjects) will be considered).

2. To evaluate in vivo, in a murine experimental model of anemia, without or with CKD, the effects of the modulation (inhibition) of iron deficiency triggers (hepcidin) and of the increase in FGF23 (HIF1alpha) on markers of cardiovascular damage. The experiments will be carried out with Wistar rats wild-type (Charles River, France) in according to the current national rules about animal well-being (BOE No. 256 of 10/25/90; Amendment Protocol to the agreement 123; 2/12/2005). Wistar rats will be fed a diet with either a normal iron content (control group, 45mg / kg diet) or low iron content (anaemic group, 5 mg / Kg diet) without or with adenine (0.2% wt/wt),which induces CKD. Diets will contain standard phosphate concentrations. Diets will begin postweaning, at 21-24 days of age, and provided ad libitum. Rats will stand on the diets for 8 wk, until the experimental end point. An additional animal group will receive intraperitoneal injections of an inhibitor of HIF1α (2-methoxyestradiol 25μg/g) (Selleckchem-Pfizer, USA) or of an inhibitor of hepcidin (AG490, 15mg/Kg) (Calbiochem), respectively. Animal diets will be obtained from Altromin (Germany). At the time of euthanasia, the investigators will collect whole blood, urine and the heart will be removed. Blood will be processed immediately to separate plasma and serum and stored at -80 ° C.2.1.1. Biochemical Parameters Serum creatinine, phosphate, and calcium will be measured by colorimetric methods (Biosystems). Serum hepcidin will be measured by ELISA (Elabsciecne). Serum vitamin D will be determined by RIA (Immunodiagnostics Systems, UK). Serum intact parathyroid hormone (iPTH), plasma C-terminal FGF23 (cFGF23), and plasma intact FGF23 (iFGF23), hepcidin concentrations will be assayed using rodent-specific ELISA kits (Immutopics, CA). Ferritin levels will be determined by mouse ELISA (Abcam, USA); serum iron will be measured spectrophotometrically (Pointe Scientific USA). BNP, myoglobin and troponin I will be evaluated by ELISA (Thermofisher scientific).

2.1. Localization of proteins in cardiac tissue through Molecular Imaging (MALDI IMAGING). The previously paraffinised hearts will be cut with a microtome to a maximum thickness of 5um and deposited in a conductive crystals previously modified with polylysine. Subsequently, a standardized dewaxing / rehydration treatment of the tissue will be performed. The tissue digestion will be carried out with trypsin deposited by sprayer and after it the most suitable matrix will be deposited to perform the analysis of the generated peptides by mass spectrometry using a mass spectrometer type MALDI-TOF /TOF (model 5800 TOF / TOF, ABSciex).

2.2. To compare in vivo, in an experimental model of anemia with and without CKD, the effect on FGF23 levels and the cardiovascular impact of different iron presentations (ferrous sulphate, ferric carboxymaltose and ferric citrate). The investigators will check the effect of different iron-based formulations (carboxymaltose ferric (Ferinject-Vifor Pharma), ferric citrate and ferrous sulphate (both of them from Sigma)) on the expression of cardiovascular markers as well as on FGF23 production.The iron restricted anemia and CKD models will be the same that were previously specified (section 2.1). The iron-based preparations will be administered intravenously. Rats will receive a single i.v. dose by tail vein injection of the corresponding iron compound (40 mg / kg body weight) or control solution (equivalent volume) at the same time every 7 days for 4 weeks. Treatment doses will be adjusted each week according to the body weight of each animal. At the time of euthanasia, the investigators will collect whole blood, which will be processed immediately and stored at -80 ° C, and will perform the biochemical analysis specified in the 2.1.1 section. Heart will be harvested, fixed in 100% ethanol, and embedded in paraffin. A histological study will be carried out in association with the pathological anatomy Service of R.S. Hospital. On the other hand, several studies describe a direct effect of PTH on FGF23 and very recent data show an increase in PTH levels after administration of Carboxymaltose. Thus, in order to assess whether the effect of Carboxymaltose on FGF23 levels is mediated through PTH, the investigators will carry out studies with Wistar rats to which we will perform a selective parathyroidectomy (PTX) and will infuse Carboxymaltose ± PTH 4X with a minipump (Alzet model 2ML4 osmotic minipump (Charles River Laboratories, Barcelona, Spain) for 14 days. The levels of PTH, FGF23i, and FGF23c will be determined.

STATISTICAL ANALYSIS. Continuous variables will be compared by Student's "t" and by Analysis of Variance (ANOVA). In the event that these variables would not follow a normal distribution, the relevant transformation of the data will be applied and nonparametric tests will be assayed. The association between categorical variables will be analyzed using the chi-square test. For the multivariate analysis of these data, the statistical procedures of Kaplan-Meier Curves analysis, conditional logistic regression and Cox regression will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Hemoglobin < 11g/dl
* Serum ferritin < 100 ng/ml or transferrin saturation index < 20%

Exclusion Criteria:

* Weight < 50 Kg or BMI < 17
* Acute bleeding > 500 ml, within 72 hours before study inclusion
* Proliferative hematologic disease. Hemochromatosis
* Active infections within 30 days before study inclusion
* Systemic inflammatory illness
* Human immunodeficiency virus (HIV), Hepatitis C virus (HCV) or Hepatitis B virus (HBV) infection
* Iron active treatment
* Blood transfusion in the last 90 days before inclusion.
* Cardiovascular hospitalization 30 days before study inclusion
* Anticoagulant treatment with coumarins
* Chronic liver disease
* Immunosuppressive therapy
* Erythropoiesis stimulating agents treatment, radiotherapy or chemiotherapy within 30 days before inclusion
* Scheduled major surgery during study period
* Pregnancy or lactation
* Drugs addiction
* Participation in others clinical trials.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Reina Sofia Hospital´s outpatients from Nephrology, Hematology an Internal Medicine services
Sampling Method: Non-Probability Sample
Enrollment: 401 (Estimated)
Dates: Start 2021-10-18 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
FGF23 on the induction of cardiovascular damage in anemia with and without CKD | 3 months
  Association between iron metabolism, FGF23 and markers of cardiovascular damage in anemia with and without CKD.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Muñoz Castañeda, MD, Principal Investigator — Maimónides Biomedical Research Institute of Córdoba
Locations (1):
- Hospital Universitario Reina Sofia, Córdoba, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Martin-Malo A, Borchard G, Fluhmann B, Mori C, Silverberg D, Jankowska EA. Differences between intravenous iron products: focus on treatment of iron deficiency in chronic heart failure patients. ESC Heart Fail. 2019 Apr;6(2):241-253. doi: 10.1002/ehf2.12400. Epub 2019 Jan 29. PMID 30694615
- [Result] Rodelo-Haad C, Santamaria R, Munoz-Castaneda JR, Pendon-Ruiz de Mier MV, Martin-Malo A, Rodriguez M. FGF23, Biomarker or Target? Toxins (Basel). 2019 Mar 22;11(3):175. doi: 10.3390/toxins11030175. PMID 30909513
- [Result] Rodriguez-Ortiz ME, Alcala-Diaz JF, Canalejo A, Torres-Pena JD, Gomez-Delgado F, Munoz-Castaneda JR, Delgado-Lista J, Rodriguez M, Lopez-Miranda J, Almaden Y. Fibroblast growth factor 23 predicts carotid atherosclerosis in individuals without kidney disease. The CORDIOPREV study. Eur J Intern Med. 2020 Apr;74:79-85. doi: 10.1016/j.ejim.2019.12.008. Epub 2019 Dec 31. PMID 31899053
- [Result] Rodriguez-Ortiz ME, Gomez-Delgado F, Arenas de Larriva AP, Canalejo A, Gomez-Luna P, Herencia C, Lopez-Moreno J, Rodriguez M, Lopez-Miranda J, Almaden Y. Serum Magnesium is associated with Carotid Atherosclerosis in patients with high cardiovascular risk (CORDIOPREV Study). Sci Rep. 2019 May 29;9(1):8013. doi: 10.1038/s41598-019-44322-z. PMID 31142774
- [Result] Rodriguez-Ortiz ME, Diaz-Tocados JM, Munoz-Castaneda JR, Herencia C, Pineda C, Martinez-Moreno JM, Montes de Oca A, Lopez-Baltanas R, Alcala-Diaz J, Ortiz A, Aguilera-Tejero E, Felsenfeld A, Rodriguez M, Almaden Y. Inflammation both increases and causes resistance to FGF23 in normal and uremic rats. Clin Sci (Lond). 2020 Jan 17;134(1):15-32. doi: 10.1042/CS20190779. PMID 31860056

DOCUMENTS (2):
  • Study Protocol (2021-12-21): https://cdn.clinicaltrials.gov/large-docs/25/NCT05356325/Prot_000.pdf
  • Informed Consent Form (2021-12-21): https://cdn.clinicaltrials.gov/large-docs/25/NCT05356325/ICF_001.pdf